CLINICAL TRIAL: NCT05495958
Title: The Efficacy and Safety of Topical Vitamin D Drop on Meibomian Gland Function in Patients With Meibomian Gland Dysfunction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14014
Record Dates: First submitted 2022-07-24; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescribe topical placebo eye drop (Placebo Comparator)
  Interventions: Drug: Topical placebo eye drop
- Prescribe topical Vitamin D eye drop (Active Comparator)
  Interventions: Drug: Topical Vitamin D eye drop

INTERVENTIONS:
Drug: Topical Vitamin D eye drop — 25 Microgram/cc or 1000 IU
  Arms: Prescribe topical Vitamin D eye drop
Drug: Topical placebo eye drop — The same-shape packed drop without vitamin D
  Arms: Prescribe topical placebo eye drop

SUMMARY:
In this randomized clinical trial, patients with Meibomian gland dysfunction aged 50 year and more will be enrolled. The Meibomian gland dysfunction diagnosis will confirmed by a cornea specialist. The enrolled patients will be randomly allocated to the treatment and placebo group. The patients in treatment group will receive topical vitamin D every 6 hours daily (25 Microgram/cc or 1000 IU). The control group will receive the same-shape packed drop without vitamin D. The patients in both group will receive the conventional treatment including hot compress and shampoo scrub.

The primary outcome is the change in Ocular surface disease index and 5-Item Dry Eye Questionnaire score assessed before the topical treatment and every one-months until 3 months. The secondary outcome measures are Tear breakup time, Schirmer test, Corneal fluorescein staining, Meibomian gland expressibility.

The grader and the patients will blind to the study group.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 50 years old and suffering from dry eye caused by meibomian gland dysfunction.

Exclusion Criteria:

* Patients with Vitamin D deficiency
* Patients taking Vitamin D systemic Supplementation
* Patient with prior ocular surgeries within previous 6 months.
* Patient with other causes of dry eye, such as aqueous tear deficiency or ocular surface disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index score | 3 months
  The standard questionnaires.

SECONDARY OUTCOMES:
Tear breakup time (TBUT) | 3 months
  time between fluorescein staining of the cul de sac and appearing dry island on the cornea
schirmer1 | 3 months
  Millimeter of the standard strip wetting by tear of the patient
Fluorescein staining test | 3 months
  The number of fluorescein stained points on the cornea & conjunctiva based on Oxford classification score

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research center, Tehran, Iran